CLINICAL TRIAL: NCT00469144
Title: A Randomized Study of Once Daily IV Busulfan With Fludarabine With Hemopoietic Stem Cell Transplantation for Acute Myelogenous Leukemia (AML) and Myelodysplastic Syndrome (MDS)
Brief Title: IV Busulfan With Allo-BMT: Study for Patients With Acute Myelogenous Leukemia and Myelodysplastic Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005-0366; NCI-2012-01475 (Registry Identifier: NCI CTRP); CA55164 (Other: NCI)
Record Dates: First submitted 2007-05-03; First posted 2007-05-04 (Estimated); Results first posted 2021-01-19 (Actual); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Myelodysplastic Syndrome; Leukemia; Acute Myeloid Leukemia
Keywords: Stem Cell Transplantation; Leukemia; Busulfan; Fludarabine; MDS; AML
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia; Leukemia, Myeloid, Acute | interventions — Busulfan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fixed-Dose Busulfan + Fludarabine (Experimental): Busulfan Fixed Dose = 130 mg/m^2 IV Daily Over Three Hours x 4 Days. Fludarabine 40 mg/m^2 IV Daily Over 1 Hour x 4 Days.
  Interventions: Drug: Busulfan; Drug: Fludarabine
- Adjusted Dose Busulfan + Fludarabine (Experimental): Busulfan Adjusted Dose = 32 mg/m^2 IV Over 2 Hours Test Dose x 1 Day. Fludarabine 40 mg/m^2 IV Daily Over 1 Hour x 4 Days.
  Interventions: Drug: Busulfan; Drug: Fludarabine

INTERVENTIONS:
Drug: Busulfan — Fixed Dose = 130 mg/m^2 IV Daily Over Three Hours x 4 Days.
  Adjusted Dose = 32 mg/m^2 IV Over 2 Hours Test Dose x 1 Day.
  Proceeding dosage level determined by pharmacokinetic studies to achieve a daily area under curve (AUC) of 6,000 microMol-min ± 10%.
Drug: Fludarabine — 40 mg/m^2 IV Daily Over 1 Hour x 4 Days

SUMMARY:
The goal of this clinical research study is to learn if giving busulfan in a dose based on blood levels, along with a fixed (unchanging) dose of fludarabine, is more effective and causes fewer side effects for AML or myelodysplastic syndrome patients than the standard method of giving a fixed busulfan dose based on body size, along with a fixed dose of fludarabine. The safety of dosing based on blood levels will also be studied.

DETAILED DESCRIPTION:
Busulfan is a chemotherapy drug that kills cancer cells by binding to DNA, and is commonly used in stem cell transplantation. Fludarabine is an antimetabolite drug which has anti-leukemia and immunosuppressive effects.

If you are eligible to take part in this study, you will be randomly assigned (as in the toss of a coin) to 1 of 2 study groups. One group will receive a fixed dose of busulfan, while the other group will receive an adjusted dose of busulfan based on blood levels of the drug. Both groups will receive fludarabine treatment as well as a stem cell transplant.

Patients in the adjusted-dose group will first receive a low-level "test" dose of busulfan to check how their blood levels change over time; this information will be used to decide the next dose needed to reach the target blood level that matches your body size. Patients in the fixed-dose group will receive a fixed dose of busulfan without the test dose. If you are assigned to the fixed-dose group, this measurement will only affect your dose level if you have an unusually high or low drug level in your blood. Patients in both groups will have a total of about 20 teaspoons (less than 7 tablespoons) of blood drawn over time to check their busulfan blood levels following one or more of the busulfan treatments.

About 11 samples of blood will be drawn to check your blood levels of busulfan over time following the test dose and the first high-dose busulfan treatment; each sample is about 1 teaspoon of blood. A heparin lock will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for these blood level tests to be performed for technical or scheduling reasons, you will receive the standard fixed dose.

Both groups of patients receive fludarabine through a central venous catheter (CVC--a small tube inserted into one of your major veins, usually in the chest or shoulder blade) over 1 hour, once a day, for 4 days. After each dose of fludarabine, the high-dose Busulfan will be infused through the CVC over 3 hours. These drugs are given to try to kill malignant cells and suppress your immune system in order to reduce the risk of stem cell transplant rejection. If you are going to be receiving a transplant from an HLA-type-nonidentical or unrelated donor, you will also receive Thymoglobulin (ATG) over 4 hours on the 3 days prior to the transplant to further suppress your immune system.

After 2 days of rest, the allogeneic stem cells (bone marrow or peripheral blood stem cells) will then be given intravenously (IV--through a needle in your vein). You will receive the drug G-CSF (Neupogen) as an injection under the skin daily starting 1 week after the transplant until your blood cell levels return to normal.

Patients usually remain in the hospital for about 4 weeks after stem cell transplantation. After you are released from the hospital, you will continue as an outpatient in the hospital area to be monitored for infections and transplant-related complications for a minimum of 100 days after the transplant.

Patients who previously had leukemia involvement in the nervous system may need to receive spinal taps, with injection of cytosine arabinoside and hydrocortisone, several times over the year after transplantation to try to keep the leukemia from coming back.

You will undergo blood tests and bone marrow biopsies at 3, 6, and 12 months after the transplant, to check if the disease is in remission. Your health status will be followed along with their local physician to find out if the leukemia or myelodysplastic syndrome comes back, as well as to check the length of your survival.

This is an investigational study. All of the drugs used in this study are approved by the FDA for treatment of cancer. Up to 230 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Acute myeloid leukemia past first remission, in first or subsequent relapse, in first remission (cytogenetics other than t(8;21, inv 16, t(15;17)) or induction failures. Only myeloid leukemia but not biphenotypic leukemia is allowed on this study.
2. Myelodysplastic syndromes with intermediate or high risk International Prognostic Scoring System score
3. Patient has not been administered any other systemic chemotherapeutic drug (including Mylotarg) within 21 days prior to trial enrollment (BMT Day -7 or day -9 for the test-dose arm of the study). Hydroxyurea is permitted if indicated to control induction refractory disease, and IT chemotherapy is allowed if indicated as maintenance treatment for previously diagnosed leptomeningeal disease, that has been in remission for at least 3 months prior to enrollment on this study).
4. No active infection. Protocol PI will be final arbiter if there is uncertainty regarding whether a previous infection is resolved.
5. age <=65
6. Patients must have a matched related or unrelated donor willing to donate. A donor who is HLA identical or mismatched in 1 locus on Class I [HLA, A or B], or molecularly mismatched in 1 locus on Class II [HLA, DR or DQ] is also acceptable.
7. ZUBROD performance status <2
8. Life expectancy is not severely limited by concomitant illness and expected to be >12 weeks.
9. Left ventricular ejection fraction >45% No uncontrolled arrhythmias or symptomatic cardiac disease.
10. No symptomatic pulmonary disease. Forced expiratory volume at one second (FEV1), forced vital capacity (FVC) and diffusion capacity of lung for carbon monoxide (DLCO) >/= 50% of expected corrected for hemoglobin. In patients </= 7 years pulmonary function will be assessed per pediatric BMT routine
11. Serum creatinine </= 1.5 mg%.
12. Serum glutamate pyruvate transaminase (SGPT) </= 200 IU/ml, serum bilirubin and alkaline phosphatase within accepted laboratory standard normal limits or considered not clinically significant. No evidence of chronic active hepatitis or cirrhosis. If positive hepatitis serology, discuss with Study Chairman and consider liver biopsy.
13. No effusion or ascites >1L prior to drainage.
14. HIV-negative.
15. Female patient is not pregnant (negative B-human chorionic gonadotropin (HCG) pregnancy test in all women of child-bearing-potential in accordance with departmental routine).
16. Patient or patient's legal representative, parent(s) or guardian able to sign informed consent.
17. No prior autologous stem cell transplants

Exclusion Criteria:

1) None.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2005-06; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard E. Champlin, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: June 28, 2005 to May 12, 2011. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: A total of 233 participants were enrolled, out of which 8 participants withdrew from study prior to treatment and are not evaluable on protocol.
Groups:
- Fixed-Dose Busulfan + Fludarabine: Busulfan Fixed Dose = 130 mg/m^2 intravenous (IV) Daily Over Three Hours x 4 Days. Fludarabine 40 mg/m^2 IV Daily Over 1 Hour x 4 Days.
- Adjusted Dose Busulfan + Fludarabine: Busulfan Adjusted Dose = 32 mg/m^2 IV Over 2 Hours Test Dose x 1 Day. Fludarabine 40 mg/m^2 IV Daily Over 1 Hour x 4 Days.
  Adjusted Dose = 32 mg/m^2 IV Over 2 Hours Test Dose x 1 Day; Proceeding dosage level determined by pharmacokinetic studies to achieve a daily area under curve (AUC) of 6,000 microMol-min ± 10%.
Period: Overall Study
Arm/Group | Fixed-Dose Busulfan + Fludarabine | Adjusted Dose Busulfan + Fludarabine
Started | 114 (Eight assigned to Fixed Dose without randomization.) | 111
Completed | 108 | 105
Not Completed | 6 | 6
Not completed — Death | 0 | 1
Not completed — No Response | 5 | 5
Not completed — Progressive Disease | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed-Dose Busulfan + Fludarabine | Adjusted Dose Busulfan + Fludarabine | Total
Number analyzed (Participants) | 114 | 111 | 225
Age, Continuous [Median (Full Range); unit: years] | 52 [14 to 66] | 50 [14 to 65] | 50 [14 to 66]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 56 | 111
  Male | 59 | 55 | 114
Region of Enrollment [Number; unit: participants]
  United States | 114 | 111 | 225

OUTCOME MEASURES:

1. Primary Outcome: Treatment-related Mortality (TRM)
Description: Time to failure (TTF) defined as either disease recurrence or death, from the time of bone marrow transplant (BMT) and reported as TRM at 100 days and 1 year.
  Treatment period defined as BMT Day -9 for patients treated on the PK-guided treatment arm, and day -7 for patients receiving the fixed-dose busulfan treatment through BMT Day +28. The post study surveillance period is defined as BMT Day +29 through BMT Day +100. Bone marrow aspirate with cytogenetics at approximately one (1) month and three (3) months, or as clinically indicated.
  Response Criteria is measured by the bone marrow aspirate to determine it has leukemic blast. Bone marrow blast less than 5% is considered to be a complete response.
Time Frame: From transplant at Day 0 to Day 100 and 1 year following transplant
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Fixed-Dose: Participants in CR; Fixed Dose: Participants Not in CR: Busulfan Fixed Dose = 130 mg/m^2 intravenous (IV) Daily Over Three Hours x 4 Days. Fludarabine 40 mg/m^2 IV Daily Over 1 Hour x 4 Days.
- Adjusted Dose: Participants in CR; Adjusted Dose: Participants Not in CR: Busulfan Adjusted Dose = 32 mg/m^2 IV Over 2 Hours Test Dose x 1 Day. Fludarabine 40 mg/m^2 IV Daily Over 1 Hour x 4 Days.
  Adjusted Dose = 32 mg/m^2 IV Over 2 Hours Test Dose x 1 Day; Proceeding dosage level determined by pharmacokinetic studies to achieve a daily area under curve (AUC) of 6,000 microMol-min ± 10%.
Arm/Group | Fixed-Dose: Participants in CR | Adjusted Dose: Participants in CR | Fixed Dose: Participants Not in CR | Adjusted Dose: Participants Not in CR
Number analyzed (Participants) | 68 | 71 | 46 | 40
Percentage of Participants
  100 Days | 3 [1 to 11] | 3 [1 to 11] | 7 [2 to 20] | 3 [0.5 to 17]
  1 Year | 19 [11 to 32] | 17 [10 to 29] | 18 [10 to 34] | 3 [0.5 to 17]
Statistical Analysis 1: Comparison: Fixed-Dose: Participants in CR vs Adjusted Dose: Participants in CR; 100 Days, Between Arms: Participants in CR; Test type: Superiority or Other; p = 0.9, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Fixed Dose: Participants Not in CR vs Adjusted Dose: Participants Not in CR; 100 Days, Between Arms: Participants not in CR; Test type: Superiority or Other; p = 0.4, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Fixed-Dose: Participants in CR vs Adjusted Dose: Participants in CR; 1 Year, Between Arms: Participants in CR; Test type: Superiority or Other; p = 0.7, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Fixed Dose: Participants Not in CR vs Adjusted Dose: Participants Not in CR; 1 Year, Between Arms: Participants not in CR; Test type: Superiority or Other; p = 0.05, Wilcoxon (Mann-Whitney)

2. Primary Outcome: 3 Year Progression Free Survival
Description: PFS defined as length of time either due to disease recurrence or death, from the time of stem cell infusion (Bone marrow or PBPC) to 3 years.
  Response Criteria is measured by the bone marrow aspirate to determine it has leukemic blast. Bone marrow blast less than 5% is considered to be a complete response.
Time Frame: 3 years
Measure: Median (Full Range); unit: Days
Arm/Group | Fixed-Dose Busulfan + Fludarabine | Adjusted Dose Busulfan + Fludarabine
Number analyzed (Participants) | 114 | 111
Days | 42 [32 to 52] | 56 [45 to 66]

ADVERSE EVENTS:
Time Frame: Adverse events collected from BMT Day -7 through BMT Day +28 or the day of discharge from the in-patient unit and post-study surveillance from initial discharge to BMT Day +100. The end of active treatment is the day of the allogeneic stem cell infusion.
Description: Overall AE collection period: July 21, 2005 to October 27, 2014.
Arm/Group | Fixed-Dose Busulfan + Fludarabine | Adjusted Dose Busulfan + Fludarabine
Serious Adverse Events (participants affected / at risk) | 2/114 | 3/111
Other Adverse Events (participants affected / at risk) | 29/114 | 26/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed-Dose Busulfan + Fludarabine (N=114) | Adjusted Dose Busulfan + Fludarabine (N=111)
Death (General disorders) | 1 (1) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Due to Pneumonia/Septic Shock
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — Due to Diffuse Alveolar Hemorrhage
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fixed-Dose Busulfan + Fludarabine (N=114) | Adjusted Dose Busulfan + Fludarabine (N=111)
Chronic Oral GvHD (Gastrointestinal disorders) | 2 (2) | 1 (1)
Renal Insufficiency (Renal and urinary disorders) | 1 (1) | 0 (0) — Due to antibiotics/Tacrolimus
Beta Hemolytic Streptococcus Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcus Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Syncytial Virus Upper Respiratory Infection (Infections and infestations) | 1 (1) | 2 (2)
Methicillin-Resistant Staphylococcus Aureus Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Influenza A Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Chronic Ocular GvHD (Eye disorders) | 3 (3) | 1 (1)
Chronic Lung GvHD (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic Vaginal GvHD (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Chronic Skin GvHD (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Ocular GvHD (Eye disorders) | 1 (1) | 3 (3)
Infection (Infections and infestations) | 10 (11) | 5 (5)
Esophageal Dysmotility (Gastrointestinal disorders) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Liver GvHD (Hepatobiliary disorders) | 3 (3) | 2 (2)
Oral GvHD (Gastrointestinal disorders) | 2 (2) | 2 (2)
Skin GvHD (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Hemorrhagic Cystitis (Renal and urinary disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
GI GvHD (Gastrointestinal disorders) | 1 (1) | 1 (1)
Blurry Vision (Eye disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Vascular disorders) | 0 (0) | 1 (1)
Vagina GvHD (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Lung GvHD (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bilirubin (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Autoimmune Hemolytic Anemia (Immune system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Engraftment Syndrome (Surgical and medical procedures) | 1 (1) | 1 (1)
Upper GI GvHD (Gastrointestinal disorders) | 0 (0) | 1 (1)
BK Virus (Infections and infestations) | 0 (0) | 1 (1)
Aspergillus Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Herpes Simplex Virus (Infections and infestations) | 1 (1) | 1 (1)
Influenza B Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus Reactivation (Infections and infestations) | 1 (1) | 2 (2)
Micrococcus Line Infection (Infections and infestations) | 0 (0) | 1 (1)
Parainfluenza Upper Respiratory Infection (Infections and infestations) | 0 (0) | 1 (1)
Pseudomonas Aeruginosa/Enterococcus Urinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Clostridum Difficile (Infections and infestations) | 0 (0) | 1 (1)
Enterococcus Faecalis Line Infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes Simplex Virus Esophagitis (Infections and infestations) | 0 (0) | 1 (1)
Alpha Hemolytic Strep Line Infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1)
Vulva GvHD (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hand-Foot Syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Parainfluenza Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Fungal Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Influenza A Virus Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Herpes Simplex Virus Oral Lesion (Infections and infestations) | 1 (1) | 0 (0)
Invasive Candida Glabrata/Fusarium Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Coli Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Branhamella Catarrhalis Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Corynebacterium/Bacil/Microbacterium Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Stenotrophomonas Maltophilia Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Epstein-Barr Virus (Infections and infestations) | 1 (1) | 0 (0)
Methicillin-Resistant Staphylococcus Aureus Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Parvovirus Viremia (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonas Aeruginosa Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Herpes Zoster Eruption (Infections and infestations) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 1 (1) | 1 (1)
Acinetobacter Calcoaceticus Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Human Herpes Virus-6 (Infections and infestations) | 2 (2) | 0 (0)
Klebsiella Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Enterococcus Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Acinetobacter Ursingii Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Parovirus B19 (Infections and infestations) | 1 (1) | 0 (0)
Stenotrophomonas (Xanthomonas) Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Bacillus Species Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Periorbital Hemorrhage (Vascular disorders) | 1 (1) | 0 (0)
Aspiration Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes